CLINICAL TRIAL: NCT06972121
Title: The Efficacy of a Digital Mindset Intervention to Improve Race Performance, Training Outcomes, and Recovery in Recreational Half Marathon Runners: A Randomized Controlled Trial
Brief Title: Digital Mindset Intervention for Half Marathon Performance
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Auckland, New Zealand (Other)
Responsible Party: Principal Investigator, Keith J Petrie, Professor, Department of Psychological Medicine, University of Auckland, New Zealand
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UAHPEC29030
Record Dates: First submitted 2025-04-14; First posted 2025-05-14 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Healthy; Exercise; Psychological Intervention
Keywords: Mindset; Exercise; Physical Activity; Sports psychology; Marathon; Performance
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mindset Intervention (Experimental): Participants in this arm are assigned to receive a digital mindset intervention designed to improve training experiences by targeting core beliefs about mindsets, and exercise symptoms such as discomfort and fatigue. This arm allows testing of the effects of mindset-focused content compared to standard training and control. Participants receive 4 brief digital modules over 9 weeks via app or email. The modules include mindset theory, reframing of physical symptoms, and race-day mental preparation.
  Interventions: Behavioral: Mindset Intervention
- Marathon Performance Training (Active Comparator): Participants in this arm are assigned to receive standard half-marathon performance training content. This arm serves as an attentional control, allowing comparison with the mindset intervention arm. Participants receive 4 brief digital modules over 9 weeks via app or email. The modules are based on publicly available running guidance and do not include any mindset-related material.
  Interventions: Behavioral: Marathon Performance Training
- Control (No Intervention): Participants in the control group will not receive any digital training or mindset content during the study period. They will continue their usual preparation for the half-marathon without additional input from the research team. This group serves as a no-intervention comparator to assess the added effects of both the mindset intervention and the marathon performance training content.

INTERVENTIONS:
Behavioral: Mindset Intervention — The mindset intervention includes 4 brief digital modules over 9 weeks (once every 3 weeks) via app or email, prior to the half-marathon race. The content introduces meta-mindsets (beliefs about how mindsets shape experiences and outcomes) and reframes non-severe physical symptoms (e.g., muscle soreness, fatigue) as signs of physiological adaptation. Modules cover: (1) what mindsets are and how they affect performance; (2) how to interpret normal training symptoms as positive signals; (3) how to maintain adaptive mindsets during peak training; and (4) race-day mindset preparation. Each module includes brief text, visuals, and reflection questions and takes approximately five minutes to complete.
  Arms: Mindset Intervention
Behavioral: Marathon Performance Training — The marathon performance training intervention includes 4 brief digital modules over 9 weeks (once every 3 weeks) via app or email, prior to the half-marathon race. Content is based on publicly available half-marathon training guidance and excludes any mindset-related material. Modules cover: (1) setting race goals and structuring training plans; (2) training tips and best practices (e.g., pacing, injury prevention); (3) navigating peak training periods (e.g., distance increases, rest and recovery); and (4) practical race-day preparation strategies (e.g., pacing, fueling, warm-up routines). Each module includes concise text, visuals, and actionable tips designed to take approximately five minutes to complete.
  Arms: Marathon Performance Training

SUMMARY:
The goal of this randomized controlled trial is to test whether a brief digital mindset training program can improve performance among recreational runners training for a half marathon in New Zealand in 2025. The study will recruit healthy adult participants who are registered for an upcoming half-marathon event.

The study aims to answer two main questions:

1. Does the mindset training program - designed to reframe common physical symptoms like fatigue or muscle soreness as signs of progress - help more runners complete the race and improve their official times, compared to standard training advice?
2. Does it support better training (e.g., longer peak training weeks) and faster physical recovery after the race?

Researchers will compare participants who receive the mindset training program to those who receive widely followed half-marathon training content and a group who receive no study content, to see whether the mindset training leads to better half-marathon performance and training outcomes.

Participants will:

* Complete a brief online survey at the start of the study
* Receive and engage with four pieces of digital content across nine weeks before the half-marathon race (if assigned to a training group)
* Complete a follow-up survey after the half-marathon

DETAILED DESCRIPTION:
This randomized controlled trial evaluates whether a brief digital mindset intervention can improve performance and training outcomes among recreational runners training for a half marathon. The intervention is grounded in psychological theories of mindsets, expectation, placebo effects, and effort perception, which suggest that how individuals interpret physical symptoms during exercise-such as fatigue or muscle soreness-can influence motivation, persistence, and overall outcomes.

The intervention aims to reframe mild physical symptoms experienced during training as signs of physiological adaptation rather than negative signals, helping participants develop more adaptive mindsets about effort and endurance. Intervention content includes brief digital modules that introduce the concept of meta-mindsets (beliefs about how mindsets influence experiences and outcomes) and provide applied strategies for interpreting discomfort as a normal and constructive part of the endurance training process.

The digital modules are delivered over a nine-week period leading up to the participant's half marathon and are designed to be time-efficient and accessible. To ensure comparability, participants assigned to the active control group receive parallel-format digital modules that focus on widely followed training advice, without any mindset-related material. Participants in the control group do not receive digital content during the study period. All intervention content is delivered via the Intervengine platform or email.

Participants are randomly assigned in a 1:1:1 ratio to one of three study arms. Randomization is conducted independently using a computer-generated allocation sequence. The study follows an intention-to-treat analysis approach, with additional per-protocol analyses among participants who complete the intervention and race.

Statistical analyses will include ANOVA and mixed-model approaches to assess group differences in primary and secondary outcomes over time. Missing data will be addressed using multiple imputation techniques. All eligibility criteria, outcome measures, and intervention details are specified in the relevant sections of the clinical trial registration record.

This trial contributes to a growing body of research examining scalable psychological interventions that support physical activity adherence and performance. It explores whether brief mindset-focused training can enhance endurance outcomes in real-world, non-clinical athletic contexts.

ELIGIBILITY:
Inclusion Criteria:

* Be aged 18 years or older
* Be registered to run (not walk) in a 2025 half marathon in New Zealand
* Be running their 1st, 2nd, or 3rd half marathon
* Be able to complete the half-marathon without physical assistance or aids
* Be able to read and understand English
* Have regular access to email or an internet-connected device

Exclusion Criteria:

* Have completed more than 2 half marathons in the past
* Are currently injured or unable to complete the race unassisted
* Are unable to complete online questionnaires independently
* Do not have access to a device capable of receiving digital content via app or email

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Official Race Times | At half-marathon race completion (approximately 9 weeks after intervention start)
  The primary study outcome is the official half-marathon finish time recorded for each participant (in hours, minutes, and seconds)
Race Completion | At half-marathon race completion (approximately 9 weeks after intervention start)
  Number of participants who complete a half marathon, across each study arm.

SECONDARY OUTCOMES:
Race Recovery | 1-week post-race (self-reported number of days to recover since race day)
  Number of days it took participants to feel fully recovered from their half-marathon race. For example, when fatigue and muscle pain subsided.
Peak Training Week Run Frequency | 1-week post-race (reflecting participant-identified peak training week, usually 3-4 weeks before race day)
  The number of days each participant ran during their peak training week before the half-marathon race.
  Measured with the question:
  During your peak training week, how many days did you train? (days/week)
Peak Training Week - Total Distance Run | 1-week post-race (reflecting participant-identified peak training week, usually 3-4 weeks before race day)
  The total distance (in kilometers) that each participant ran across all training runs during their peak training week prior to the half-marathon race.
  Measured with the question:
  During your peak training week, what was the total distance you ran across all your runs that week? (km)

OTHER OUTCOMES:
Adapted Body Mindset Inventory | From baseline to 1-week post-race.
  The Body Mindset Inventory - Version 2 (BMI-2), adapted for half-marathon runners.
  Assessed using 6-point Likert scale (1 = Strongly disagree, 6 = Strongly agree).
Mindset vs. Training Attribution | 1-week post-race (reflecting 9-week intervention period)
  Perceived influence of mindset vs. training schedule on race performance
  Assessed via two self-report items using 10-point Likert scales (1 = Not at all, 10 = An extreme amount):
  "How much do you think your mindset influenced your half marathon training and performance?"
  "How much do you think your training schedule influenced your half marathon performance?"
  A difference score will be calculated by subtracting the response to item 2 (training schedule) from item 1 (mindset). This score reflects the participant's relative attribution of their performance to mindset vs. training. Positive scores indicate greater perceived influence of mindset; negative scores indicate greater influence of the training schedule.
Interpretation of Exercise Symptoms as Signs of Adaptation | From baseline to 1-week post-race
  The extent to which participants interpret common sensations during challenging runs (e.g., fatigue, muscle discomfort, heavy breathing) as indicators that their body is getting stronger. Responses are collected using a 10-point visual analogue scale ranging from 1 ("not at all signs of getting stronger") to 10 ("definitely signs of getting stronger").
Belief in the Controllability of One's Mindset | From baseline to 1-week post-race
  Participants' belief in their ability to influence their mindset, even in high-stakes situations, measured using one item from the Controllable Meta-Mindset Scale: "Even in moments when it really matters, I can't do much to change my mindset." Responses are rated on a 6-point Likert scale (1 = Strongly disagree, 6 = Strongly agree).
Perceived Influence of Expectations on Performance | At baseline
  Participants' beliefs about the role of expectations in their upcoming half-marathon performance. Measured using a single item:
  "To what extent do you think your expectations will affect your half-marathon performance?", using a 6-point Likert scale (1 = Not at all, 6 = An extreme amount)
Motivation and Future Intentions | 1-week post-race
  How likely study participants are to participate in another half marathon or endurance race. Measured with 5-point Likert scale (1 = Not at all likely, 5 = Extremely likely).
Satisfaction with Race Day Performance | 1-week post-race
  How satisfied people are with their race day performance. Measured with 5-point Likert scale (1 = Not at all satisfied, 5 = Very satisfied).
Change from Previous Half-Marathon Personal Best Time | Within 15 minutes after half-marathon race completion
  Change in half-marathon race time, calculated as the difference (in minutes:seconds) between each participant's self-reported previous personal best and their official finish time in their 2025 half-marathon (for those with a prior half-marathon result).
Achievement of Half-Marathon Race Goal Time | 1-week post-race
  Did participants perform better or worse than their goal time for the half marathon. Measured via a single-item question administered post-race: "Was this time better or worse than your goal time?" Participants select one of four response options: Better; About the same; Worse; I did not have a goal time
Running-Related Injuries | Up to 16 weeks post-enrollment (assessed 1-week post-race)
  Whether participants experienced any running-related injuries, measured with a single yes/no response question. Since enrolling in this study, did you experience any running-related injuries - before, during, or after your half-marathon race? (Yes (please specify) / No)
Self-Reported Training Adherence | 1-week post-race (covering up to 15 weeks of training)
  Participants' self-reported adherence to their intended training plan in the weeks leading up to the race. Assessed via a single-item question using a 5-point Likert scale:
  "How often did you follow your planned training sessions in the weeks leading up to the race?" (1 = Rarely followed my plan, 5 = Followed my plan consistently)
Open-Text Reflections on Expectations for the Half Marathon | At baseline
  Participants are invited to provide an optional open-text response to the prompt: "What thoughts come to mind when you think about your upcoming half marathon right now?" This will be used to explore participants' anticipatory beliefs and expectations before training and intervention delivery.
Reflections on Training and Race Experience | 1-week post-race
  Participants are invited to complete two optional follow-up prompts:
  1. an open-text reflection on how their training and participation in the Mount Maunganui Half Marathon 2025 went, and
  2. a brief prompt asking them to provide two words that best describe their overall experience.
  These responses will be used to qualitatively explore participant perceptions of their training journey and race experience.
Intervention Evaluation | 1-week post-race (reflecting 9-week intervention period)
  Acceptability of the intervention content. Measured with four summed items on a 5-point Likert scale (Scale: 1 = Strongly disagree, 5 = Strongly agree).
  The digital content was clear and easy to understand. The digital content helped me perform better during my half marathon. The digital content motivated me to stay consistent with my training. The digital content helped me reframe discomfort during training and my half marathon in a helpful way.
Half-Marathon Experience Level | At baseline
  Participants' prior experience with half-marathon events. Measured using a single self-report item: "How would you describe your half-marathon experience level?" Participants select from two predefined options: (1) Beginner (training for your first half marathon) (2) Intermediate (previously completed up to 2 half marathons).
Previous Personal Best Half-Marathon Time (for Intermediate Runners) | At baseline
  Self-reported fastest half-marathon finish time to date. Participants enter their best recorded time in hours and minutes.
Current Weekly Running Frequency | At baseline
  How often participants currently run each week. Measured with a single self-report item: "How many days per week do you currently run for exercise?" Options: None; 1 day; 2-3 days; 4-5 days; 6-7 days.
Average Distance of Current Runs | At baseline
  Participants' typical running distance per session. Measured using a self-report item: "What is the average distance of your current runs (in kilometers)?"
Half-Marathon Training Plan Status | At baseline
  Whether participants are following a structured training plan for their upcoming race. Measured with a Yes/No self-report question: "Do you have a training plan for your Half Marathon?"
Goal Time for Half-Marathon | At baseline
  Participants' target finish time for the upcoming half marathon. Measured via a self-report item: "Do you have a goal time for the half marathon?" If yes, participants specify their goal time in hours and minutes.
Typical Recovery Time After Long Runs | At baseline
  How long participants typically take to recover from a long training run. Measured with a single self-report item: "How many days do you typically take to recover from a long run?" Options: 1 day; 2 days; 3 or more days; N/A (I haven't started running yet).

CONTACTS AND LOCATIONS:
Overall Officials: Keith Petrie, Professor, Principal Investigator — University of Auckland, New Zealand
Locations (1):
- Faculty of Medical and Health Sciences, University of Auckland, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be made available due to ethical and privacy considerations outlined in the study's protocol. Participants did not provide consent for their individual-level data to be shared beyond the research team. In line with University of Auckland ethics guidelines, data sharing is limited to de-identified, aggregated results reported in publications or presentations.